CLINICAL TRIAL: NCT05950269
Title: Walking Aid and Locomotion Knowledge in Emergency Rooms (WALKER 1): Training and Provision of Walking Aids to Promote Autonomy and Mobility of Elderly People in Emergency Care - a Randomized Clinical Trial
Brief Title: Walking Aid and Locomotion Knowledge in Emergency Rooms (WALKER 1) for Elderly People
Acronym: WALKER 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVAP-NG 2999
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Mobility Limitation
Keywords: Geriatric; Life space; Walking aids; Emergency room; Clinical Trial; Mobility
MeSH Terms: conditions — Mobility Limitation; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study will be blind for the researchers involved in the post-telemonitoring assessments. Also, the data will be analyzed by a researcher who is not involved in the interventions or the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Walking aid (WA) group (Experimental): Participants will receive the walking aid and training in the use of the device.
  Interventions: Device: Walking aid; Other: Guidance on safe walking and risk of falling
- Walking aid with telemonitoring (WAT) group (Experimental): Participants will receive the walking aid and training in the use of the device associated with telemonitoring.
  Interventions: Device: Walking aid; Other: Telemonitoring; Other: Guidance on safe walking and risk of falling
- Control group (Other): Participants will receive verbal guidance and printed material.
  Interventions: Other: Guidance on safe walking and risk of falling

INTERVENTIONS:
Device: Walking aid — A physiotherapist will identify the mobility needs and will indicate the most appropriate walking aid (cane or walker).
  Arms: Walking aid (WA) group; Walking aid with telemonitoring (WAT) group
Other: Telemonitoring — Telemonitoring will occur every two weeks for three months after the emergency department discharge, through video call (about 15 minutes). On these opportunities, the importance of using mobile devices and the guidance on safe gait will be reinforced.
  Arms: Walking aid with telemonitoring (WAT) group
Other: Guidance on safe walking and risk of falling — Participants will receive verbal guidance and printed material with guidance on safe walking and fall prevention.

SUMMARY:
Older adults have higher rates of emergency department admissions when compared to their younger counterparts. Mobility is the ability to move around but also encompasses the environment and the ability to adapt to it. Walking aids can be used to improve mobility and prevent falls. According to international guidelines, they must be available in Geriatric Emergency Department. This study aims to evaluate the effectiveness of a program of training and provision of walking aids (WA), associated or not with telemonitoring, on mobility, quality of life, fear of falling, and risk of falls up to 3 months in older adults cared for in an emergency department.

DETAILED DESCRIPTION:
A randomized clinical trial will be carried out in the emergency department of Hospital Sírio-Libanês. Participants will be randomized and allocated into three intervention groups, as follows: A) Walking aid group; B) Walking aid and telemonitoring group; C) Control group. Patients will undergo a baseline evaluation encompassing sociodemographic and clinical data, mobility in life spaces (Life Space Assessment), gait speed, muscle strength, functionality (Barthel Index, Katz index, and Lawton-Brody Scale), quality of life (Euro Quality of Life Instrument-5D), fear of falling (Falls Efficacy Scale International), history of falls, cognition (10-Point Cognitive Screener) and mood (15-point Geriatric Depression Scale) before the intervention. Gait time and fear of falling will be assessed again after the intervention. Finally, mobility in life spaces, functionality, quality of life, fear of falling, history of falls, cognition, and mood will be assessed 3 months after discharge from the geriatric emergency department through a telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* Admitted to the Geriatric Emergency Department of Hospital Sírio-Libanês
* Willing and able to give informed consent
* Least one of the following for indication and training of mobility aids: reduction of postural instability; improvement of motor control; increase of somatosensory feedback; reduction of biomechanical overload; safe promotion of autonomy; fall history (in the last six months).

Exclusion Criteria:

* Altered level of conscience
* need for supplemental oxygen (≥3L/min)
* respiratory distress
* hemodynamic instability
* postural instability with a tendency to fall backward
* cognitive impairment that limits the use of walking aids
* hospitalization after Emergency Department evaluation
* Delirium

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 153 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Life-Space Assessment (LSA) | At baseline and after completion of the 3 and 6 months intervention to assess change
  LSA is a scale which allows the characterization of mobility in life-spaces specifically frequency, need for mobility aids and the help of third party in the last 4 weeks
Falls Efficacy Scale International (FES-I) | At baseline, immediately after the intervention and after completion of the 3 and 6 months intervention to assess change
  Assesses fear of falling

SECONDARY OUTCOMES:
Timed Up and Go test (TUG) | At baseline and immediately after the intervention
  TUG evaluate mobility, balance, gait, and risk of falling
One-minute sit-to-stand test | At baseline and after completion of the 3 and 6 months intervention to assess change
  Functional capacity assessment by sit and stand completely in a chair (as often as possible during 1 minute)
Katz index | At baseline and after completion of the 3 and 6 months intervention to assess change
  Katz index is a scale which evaluate basic activities of daily living
Barthel index | At baseline and after completion of the 3 and 6 months intervention to assess change
  Barthel index is a scale which evaluates the autonomy for self-care, in addition to mobility
Lawton-Brody scale | At baseline and after completion of the 3 and 6 months intervention to assess change
  Lawton-Brody scale evaluate Instrumental activities of daily living
Euro Quality of Life Instrument-5D (EQ-5D) | At baseline and after completion of the 3 and 6 months intervention to assess change
  EQ-5D evaluate quality of life in five health dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and self-rated health on a visual analog scale
Geriatric Depression Scale (GDS-15) | At baseline and after completion of the 3 and 6 months intervention to assess change
  Assesses mood disorders
10-Point Cognitive Screener (10-CS) | At baseline and after completion of the 3 and 6 months intervention to assess change
  10-CS consists of a brief cognitive screening which evaluate temporal orientation, verbal fluency and three-word recall
Fall History | At baseline and after completion of the 3 and 6 months intervention to assess change
  Fall history evaluate occurrence of falls (including data location, associated injuries, need for special care after the fall) and the total number of falls

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio Libanês, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Kennedy RE, Williams CP, Sawyer P, Lo AX, Connelly K, Nassel A, Brown CJ. Life-Space Predicts Health Care Utilization in Community-Dwelling Older Adults. J Aging Health. 2019 Feb;31(2):280-292. doi: 10.1177/0898264317730487. Epub 2017 Sep 14. PMID 29254407
- [Background] Shimada H, Sawyer P, Harada K, Kaneya S, Nihei K, Asakawa Y, Yoshii C, Hagiwara A, Furuna T, Ishizaki T. Predictive validity of the classification schema for functional mobility tests in instrumental activities of daily living decline among older adults. Arch Phys Med Rehabil. 2010 Feb;91(2):241-6. doi: 10.1016/j.apmr.2009.10.027. PMID 20159128
- [Background] Brown CJ, Kennedy RE, Lo AX, Williams CP, Sawyer P. Impact of Emergency Department Visits and Hospitalization on Mobility Among Community-Dwelling Older Adults. Am J Med. 2016 Oct;129(10):1124.e9-1124.e15. doi: 10.1016/j.amjmed.2016.05.016. Epub 2016 Jun 8. PMID 27288857
- [Background] van den Berg N, Schumann M, Kraft K, Hoffmann W. Telemedicine and telecare for older patients--a systematic review. Maturitas. 2012 Oct;73(2):94-114. doi: 10.1016/j.maturitas.2012.06.010. Epub 2012 Jul 17. PMID 22809497
- [Background] Bateni H, Maki BE. Assistive devices for balance and mobility: benefits, demands, and adverse consequences. Arch Phys Med Rehabil. 2005 Jan;86(1):134-45. doi: 10.1016/j.apmr.2004.04.023. PMID 15641004
- [Derived] Polesel FS, Denadai S, Morinaga CV, Madalena IC, Aliberti MJR, Henrique EA, de Andrade-Junior MC, Nucci RAB, Yamaguti WP, Curiati PK, Righetti RF. Walking Aids and Locomotion Training in the Emergency Department: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2544535. doi: 10.1001/jamanetworkopen.2025.44535. PMID 41269694
- [Derived] Polesel FS, Denadai S, Aliberti MJR, Morinaga CV, Andrade-Junior MC, Madalena IC, Yamaguti WP, Curiati PK, Righetti RF. Training and provision of mobility aids to promote autonomy and mobility of older patients in a geriatric emergency department: A protocol for a randomized controlled trial. PLoS One. 2024 Jul 31;19(7):e0304397. doi: 10.1371/journal.pone.0304397. eCollection 2024. PMID 39083494